CLINICAL TRIAL: NCT01217502
Title: Self-management for Dual Sensory Impaired Older People and Their Caregivers: an Effective Approach?
Brief Title: Self-management for Dual Sensory Impaired
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Kalorama 1
Record Dates: First submitted 2010-09-13; First posted 2010-10-08 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Hearing Loss; Low Vision
Keywords: Aged; Homes for the aged; Self management; Personal autonomy; Disease management; Self efficacy; Participation
MeSH Terms: conditions — Hearing Loss; Vision, Low | interventions — Self-Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Self management (Experimental)
  Interventions: Behavioral: Self management program

INTERVENTIONS:
Behavioral: Self management program — Professional caregivers will be trained in offering a self management program to aged persons with a dual sensory impairment. Duration of the program: 6 months
  Other Names: Empowerment
Behavioral: self management program — Learning and practicing skills necessary to carry on an active and emotionally satisfying life in the face of the dual sensory impairment
  Other Names: self efficacy

SUMMARY:
This study aims to determine the effectiveness of a self-management program for elderly with an acquired and concurrent hearing and visual impairment due to age-related disease processes.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of hearing loss and low vision
* at least one sensory loss acquired after the age of 55
* living in a home for the elderly

Exclusion Criteria:

* congenital deaf persons
* a dual sensory loss before the age of 55

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Participation in social, leisure and communicative activities. | 6 months
  2 outcome measures will be used:
  * Activity Card Sort (Baum & Edwards 2001): change from baseline in leisure activities and social contacts at 6 months
  * Hearing Handicap Questionnaire (Gatehouse & Noble 2004): change from baseline in communicative contacts at 6 months

SECONDARY OUTCOMES:
work satisfaction professional caregivers | 6 months
Depressive feelings | 6 months
Autonomy. | 6 months
  Outcome measure: 9-item Patient Autonomy Questionnaire (Vernooij-Dassen & Osse 2005): change from baseline in dependency, losing control, and limitation of activities at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: M. Vernooij-Dassen, Prof. dr., Study Chair — Radboud University Nijmegen Medical Centre, The Netherlands
Locations (4):
- Netherlands (4):
  - Foundation Riethorst Stromenland, Geertruidenberg, Gelderland
  - Foundation Zorggroep Noord-Limburg, Herkenbosch, Limburg
  - Maasduinen Foundation, Kaatsheuvel, North Brabant
  - Zorgbalans Foundation, Haarlem, North Holland

REFERENCES:
- [Derived] Roets-Merken LM, Zuidema SU, Vernooij-Dassen MJFJ, Teerenstra S, Hermsen PGJM, Kempen GIJM, Graff MJL. Effectiveness of a nurse-supported self-management programme for dual sensory impaired older adults in long-term care: a cluster randomised controlled trial. BMJ Open. 2018 Jan 24;8(1):e016674. doi: 10.1136/bmjopen-2017-016674. PMID 29371264
- [Derived] Roets-Merken LM, Vernooij-Dassen MJ, Zuidema SU, Dees MK, Hermsen PG, Kempen GI, Graff MJ. Evaluation of nurses' changing perceptions when trained to implement a self-management programme for dual sensory impaired older adults in long-term care: a qualitative study. BMJ Open. 2016 Nov 17;6(11):e013122. doi: 10.1136/bmjopen-2016-013122. PMID 27856482
- [Derived] Roets-Merken LM, Graff MJ, Zuidema SU, Hermsen PG, Teerenstra S, Kempen GI, Vernooij-Dassen MJ. Effectiveness of a self-management program for dual sensory impaired seniors in aged care settings: study protocol for a cluster randomized controlled trial. Trials. 2013 Oct 7;14:321. doi: 10.1186/1745-6215-14-321. PMID 24099315